CLINICAL TRIAL: NCT02932059
Title: Evaluation of Metamemory Using a Semantic Construction Strategy in Patients With Schizophrenia
Acronym: Metamemory 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: LAPSCO, Psychology University, Blaise Pascal University, Clermont-Ferrand. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHU-0280; 2016-A00944-47 (Other: 2016-A00944-47)
Record Dates: First submitted 2016-10-04; First posted 2016-10-13 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2016-10

CONDITIONS: Schizophrenia; Aging
Keywords: Metamemory; Schizophrenia; Aging; Learning; Judgement of learning; Sentence construction strategy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adult schizophrenic patients (18-45 years) (Experimental): 4 groups formed by the case-control study in two age strata
  Interventions: Behavioral: Metamemory
- Aged patients with schizophrenia (≥ 55 years) (Experimental): 4 groups formed by the case-control study in two age strata
  Interventions: Behavioral: Metamemory
- Adults controls (18-45 years) (Experimental): 4 groups formed by the case-control study in two age strata
  Interventions: Behavioral: Metamemory
- Aged Controls (≥ 55 years) (Experimental): 4 groups formed by the case-control study in two age strata
  Interventions: Behavioral: Metamemory

INTERVENTIONS:
Behavioral: Metamemory — Metamemory evaluation using a sentence construction strategy

SUMMARY:
The purpose of this study is to determine the respective roles of aging and schizophrenia in the regulation of metamemory using a sentence construction strategy. 4 groups will be necessary to comparison:

Adult patients (18-45 years) Adult controls (18-45 years) Aged patients (≥ 55 years) Aged controls (≥ 55 years)

The effects of age and the disease could lead to interaction in regulating metamemory. The effect of age would be aggravated by the disease.

DETAILED DESCRIPTION:
Metamemory measurement

* Objective: Measurement of monitoring and control capabilities, and relations between these two abilities when learning of word pairs.
* Description: The hardware consists of two lists of 30 pairs of French words, each pair of words being composed of a word index and a target word (names of concrete objects). Among the 60 word pairs, 30 are strongly associated items (or easy items, the other 30 being weakly associated or difficult items.

In front of a computer screen, each participant is subjected to a first learning test in which 30 pairs of words appear one by one on the screen. Participants have the option to control the time of presentation of each pair of words. After a retention time of 4 minutes of information devoted to nonverbal distractive task, follows an evaluation phase of deferred judgments of learning (JOL time), where for each pair of words studied, the word index is presented without the target word. Participants must then assess a learning judgment for each pair of words, that is to say they have to estimate, on a 5-point scale, their ability to remember later the target word in the presentation the index word. This JOL (judgments of learning ) assessment phase is immediately followed by cued recall test.

For the second learning test (30 other word pair), the steps are identical. Prior to this second learning, building instruction of a phrase with two words to learn is proposed. Participants are trained on 5 pairs of words. The study concludes with a question phase, during which participants give their impressions of the experience, describe the learning strategies they used and generally consider their ability mnemonic during daily tasks.

ELIGIBILITY:
Inclusion Criteria:

* For both:
* MMSE score greater than or equal to,

  * 22 if no grade
  * 23 if study certificate or CAP or college without patent
  * 25 if patent or school without the tray
  * 26 or more when bin
* IQ ≥ 75 (fNART)
* Age: between 18 and 45 years for adults, and 55 and older for older,

For patients :

* DSM-5 criteria of schizophrenia
* Adult patients (<45 years) will be matched to elderly patients (> 55 years) gender and IQ,
* Patients followed as outpatients,
* Age of onset of the disease less than 40 years,
* Patients whose disease has stabilized: no changes psychotropic treatment for at least 1 month
* Not more of a benzodiazepine,
* Patients on protection of justice or not,

For controls :

* - Matched for sex to patient
* Age-matched (+/- 3 years) to patient
* Matched for IQ (score fNART +/- 10%) to patients

Exclusion Criteria:

* For patients :
* Any other comorbid psychiatric diagnosis of Axis I DSM-5
* Extrapyramidal syndrome or tardive dyskinesia (AIMS score <2 BARS score <2 and score Simpson and Angus <3)
* Calgary depression scale ≥ 6
* Current or past addiction to all toxic substances (including alcohol and cannabis) except tobacco.
* Current or past use of all toxic consumption (excluding alcohol, tobacco and cannabis).
* Use of alcohol or cannabis before the age of 15 years
* Alcohol abuse in the past 6 months.
* Cannabis abuse in the past 6 months and cannabis use in the last 3 months.
* Patients with impaired vision or hearing preventing the realization of the tests.

For controls:

* Any psychiatric diagnosis according to DSM-5, including addictions (excluding tobacco)
* Score HADS Anxiety ≥ 8 and Depression ≥ 8
* SCL90R: global severity score GSI> 0.33 for women and> 0.27 for men, or score diversity PST symptoms> 18.49 for men and> 21.97 for women or score of degree of discomfort PSDI> 1.27 for men and> 1.3 for women, scoring in the subscale Psychotic Features> 0.
* Presence of a personality disorder at PDQ4 +
* Head injuries, brain injuries or diseases,
* vision or hearing problems preventing the realization of the tests.
* Current or past addiction to all toxic substances (including alcohol and cannabis) except tobacco.
* Current or past use of all toxic consumption (excluding alcohol, tobacco and cannabis).
* Long-term Anticholinergic treatment.
* Related to the first degree diagnosed with a psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
difference of judgement of learning using a 5 point scale (0%, 25%, 50%, 75%, 100%) in the sentence construction strategy | at day 1
  the 4 groups of participants formed by the case-control study in two age strata value their judgments of learning for each pair of words using a 5 point scale (0%, 25%, 50%, 75%, 100%) in the sentence construction strategy.
  Four groups are :
  * Adult schizophrenic patients (18-45 years)
  * Aged patients with schizophrenia (≥ 55 years)
  * Adults controls (18-45 years)
  * Aged controls (≥ 55 years)

SECONDARY OUTCOMES:
difference of judgement of learning using a 5 point scale (0%, 25%, 50%, 75%, 100%) between sentence construction and reading strategies. | at day 1
  the 4 groups of participants formed by the case-control study in two age strata, value their judgments of learning for each pair of words using a 5 point scale (0%, 25%, 50%, 75%, 100%) in a sentence construction strategy and in a reading strategy.
  For each group, difference between these two strategies will be compared.
  Four groups are :
  * Adult schizophrenic patients (18-45 years)
  * Aged patients with schizophrenia (≥ 55 years)
  * Adults controls (18-45 years)
  * Aged controls (≥ 55 years)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle JALENQUES, Principal Investigator — CHU Clermont-Ferrrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France